CLINICAL TRIAL: NCT00786214
Title: Treatment of Functional Dyspepsia With Acupuncture: A Randomized, Blinded, Sham Acupuncture Controlled Study
Brief Title: Treatment of Functional Dyspepsia With Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Medicine, Professor & Senior Consultant Gastroenterologist, Ho Khek Yu, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D/06/479
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; Acupuncture; Traditional Chinese Medicine
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Patients given acupuncture treatment
  Interventions: Other: Acupuncture
- Sham acupuncture (Sham Comparator): Patients given sham acupuncture treatment
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture — Patients will be stimulated at specific acupuncture points as determined for treatment of the disease by certified acupuncturists
  Arms: Acupuncture
Other: Sham acupuncture — Patients will be given sham acupuncture treatment at dummy acupuncture points
  Arms: Sham acupuncture

SUMMARY:
Functional dyspepsia (FD) is one of the most common chronic gastrointestinal disorders affecting humans. Existing therapies for FD are still far from satisfactory and new therapies are constantly being sought. Acupuncture has been used for the alleviation of functional gastrointestinal symptoms in several non-controlled studies. This study aims to investigate the therapeutic efficacy of acupuncture in patients with FD.

ELIGIBILITY:
Inclusion criteria:

- female and male patients with functional dyspepsia between the ages of ≥18 and ≤70 years. FD will be diagnosed according to the Rome-III criteria. Onset of FD symptoms should begin at least 6 months before clinical presentation and must be fulfilled for the last 3 months and his or her FD symptoms score must be of at least moderate severity.

Exclusion criteria:

* Subjects unable to give informed consent
* Pregnant or breast-feeding females or women who get pregnant midway
* Subjects who have received acupuncture treatment before
* Subjects who have had a previous gastrointestinal surgery except appendectomy and laparoscopic cholecystectomy
* Any significant past or concurrent disease or disorder which, in the opinion of the investigator, may either put subject at risk in the study, influence the results of the study or influence subject's ability to participate in the study
* Maintenance treatment with PPIs (proton pump inhibitors) and H2RAs (H2-receptor antagonists) continuously (every day) in the last 6 months prior to entry into the study
* Treatment with PPIs and H2RAs, prokinetics, antibiotics, prostaglandins or bismuth-containing compounds during the last 2 weeks prior to entry into the study
* H. pylori eradication treatment within the past 12 months before study start
* H. pylori positive patients
* Patients with bleeding diathesis
* Known or suspected hypersensitivity to acupuncture.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Resolution of symptoms | 4 weeks

SECONDARY OUTCOMES:
Health-related quality of life and hospital anxiety & depression scale | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Khek Yu Ho, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore